CLINICAL TRIAL: NCT06776913
Title: Randomized Controlled Trial Comparing Adult to Pediatric Colonoscope in Obese Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cleveland Clinic Florida (Other)
Responsible Party: Principal Investigator, Asad Ur Rahman, Fnu, Medical Director, Inflammatory Bowel Disease Center, Cleveland Clinic Florida
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 24-891
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Obesity (Body Mass Index &Amp;Amp;gt;30 kg/m2); Screening Colonoscopy
Keywords: obesity; Screening Colonoscopy
MeSH Terms: conditions — Obesity | interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Adult Colonoscope (Active Comparator): Adult colonoscope
  Interventions: Device: Colonoscopy
- Pediatric Colonoscope (Active Comparator): Pediatric colonoscope
  Interventions: Device: Colonoscopy

INTERVENTIONS:
Device: Colonoscopy — Standard Colonoscopy with photo documentation and the recording of procedure timing.

SUMMARY:
The goal of this study is to test which colonoscope works best in people who are above a certain body mass index. Currently, both pediatric and adult colonoscopes are accepted as standard treatments in colonoscopies. Endoscopist pick which one to use based on personal preference and what is available.

ELIGIBILITY:
Inclusion Criteria:

* BMI greater than 30
* Screening and surveillance colonoscopy

Exclusion Criteria:

* Colon surgery
* Therapeutic colonoscopy
* Inflammatory bowel disease
* Terminated procedure due to stool burden, stenosis, or obstructive mass.
* Colonoscopy for anemia
* History of incomplete colonoscopy due to technical difficulties

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
Composite of reaching the cecum in less than 10 minutes without changing the scope type. | During Surgery
  The outcome aims to measure the difficult colonoscope which is defined as either not reaching the cecum, needing more than 10 minutes, or the need to exchange to a different device.

SECONDARY OUTCOMES:
Cecal intubation rate (CIR) | During Surgery
  The percentage of successful advancement of colonoscope to the cecum.
Terminal ileum intubation rate (TIIR) | During Surgery
  The percentage of successful advancement of colonoscope to the terminal ileum.
Insertion time (IT) | During Surgery
  Time from insertion to cecum.
Withdrawal time | During Surgery
  Time from terminal ileum picture or last cecal picture to rectal picture. Subtract 1 min per each intervention (polypectomy, cauterization...)
Ancillary maneuvers used | During Surgery
  Using ancillary maneuvers during colonoscopy (position change, pressure application, increase stiffness, etc...)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Weston, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided